CLINICAL TRIAL: NCT03515278
Title: Effect of Ultrasound-guided Suprascapular Nerve Block Versus Intra-articular Corticosteroid Injection for Frozen Shoulder: a Randomized Control Trial
Brief Title: Effect of Ultrasound-guided Suprascapular Nerve Block Versus Intra-articular Corticosteroid Injection for Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170915R; 2018SKHADR029 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2018-04-13; First posted 2018-05-03 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-01

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; adhesive capsulitis; ultrasound-guided intervention; suprascapular nerve block; intra-articular injection
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suprascapular nerve block (SCNB) group (Experimental): SCNB with physiotherapy. Suprascapular nerve block: Ultrasound-guided SCNB by 3 c.c. 1% lidocaine with 20mg triamcinolone.
  Physiotherapy: The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise. (stretching, mobilization and ROM exercise, and strengthening)
  Interventions: Procedure: SCNB group
- intra-articular corticosteroid injection (IACI) group (Active Comparator): IACI with physiotherapy. Intra-articular steroid Injections: Receive intra-articular corticosteroid injection.Ultrasound-guided IACI with 3c.c. 1% lidocaine and 20mg triamcinolone.
  Physiotherapy: The physiotherapy program includes physical modalities (heat therapy and electric therapy) and therapeutic exercise. (stretching, mobilization and ROM exercise, and strengthening)
  Interventions: Procedure: IACI group

INTERVENTIONS:
Procedure: SCNB group — IACI can provide rapid effect in pain reliving, reducing inflammation and improving ROM that could increase the compliance of exercise therapy.
  Other Names: IACI group
  Arms: suprascapular nerve block (SCNB) group
Procedure: IACI group — SCNB is a new choice for treatment of frozen shoulder.As radiology techniques advance, ultrasound-guided SCNB becomes more popular. It provides a cost and time-effective way to infiltrate the nerve accurately without injury to the nerves or vessels.
  Other Names: SCNB group
  Arms: intra-articular corticosteroid injection (IACI) group

SUMMARY:
The investigators aim to compare the effect of ultrasound-guided suprascapular nerve block and intra-articular corticosteroid injection for frozen shoulder in pain control, improvement of range of motion, quality of life, and function.

DETAILED DESCRIPTION:
The inclusion criteria is: 1. unilateral side involvement; 2. ≥50% loss of passive ROM (external rotation or abduction) in the glenohumeral joint comparing to the unaffected side; 3. duration of symptoms ≥3 months. 4. age≥ 20year old.

The exclusion criteria include: 1. ever received manipulation of the affected shoulder with/without anesthesia; 2. systemic disease, severe degeneration, or trauma involving the shoulder (ie, rheumatoid arthritis, osteoarthritis, history of injury to the labrum or articular cartilage or malignancies in the shoulder region, etc.); 3. neurologic diseases such as stroke or peripheral nerve neuropathy that have already affect the activity of shoulder; 4.pain or disorders of the cervical spine, elbow, wrist, or hand; 5.a history of drug allergy to local or corticosteroids; 6. Pregnancy or lactation; and 7. Received corticosteroids, or hyaluronic acid intra-articular injection into the affected shoulder during the preceding 4 weeks 70 participants will be randomly divided to SCNB group and IACI group. Each subject in either group will receive 2 times of injection in a two-weekly interval. After injection, each subject in either group will receive the same protocol of physiotherapy program for 2 months. Outcome measures include the SPADI, the SDQ, active and passive ROM of the affected shoulder, and SF-36. Evaluation will be performed at baseline and at 4 weeks and 12 weeks after the beginning of the treatment. Statistics will be performed after completing the patients' treatment and evaluations.

A Shapiro-Wilk test will be applied to ensure that all the calculated variables followed a normal distribution. Subsequently, a 2-by-3, 2-way mixed-model analysis of variance, which has 1 between-subject factor (group: SCNB and IACI) and 1 within-subject factor (evaluation time: pretreatment, 4 weeks after beginning treatment, and 12 weeks after the beginning of the treatment), will be performed. Pair-wise comparisons between groups will be performed using an independent t test when a significant interaction is found; otherwise, the main effects are reported. When a time effect is found, a post hoc analysis will be performed using a polynomial test to determine the trend (linear or quadratic). All significance levels are set at alpha=.05, and SPSS version 15.0a will be used for all the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. unilateral side involvement.
2. ≥50% loss of passive ROM (external rotation or abduction) in the glenohumeral joint comparing to the unaffected side.
3. duration of symptoms ≥3 months.
4. age≥ 20year old.

Exclusion Criteria:

1. ever received manipulation of the affected shoulder with/without anesthesia.
2. systemic disease, severe degeneration, or trauma involving the shoulder. (ie, rheumatoid arthritis, osteoarthritis, history of injury to the labrum or articular cartilage or malignancies in the shoulder region, etc.)
3. neurologic diseases such as stroke or peripheral nerve neuropathy that have already affect the activity of shoulder.
4. pain or disorders of the cervical spine, elbow, wrist, or hand.
5. a history of drug allergy to local or corticosteroids.
6. Pregnancy or lactation.
7. Received corticosteroids, or hyaluronic acid intra-articular injection into the affected shoulder during the preceding 4 weeks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change of scores of the Shoulder Pain and Disability Index (SPADI) | baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The total SPADI score, which ranges between 0 and 100, is calculated by averaging the scores from the pain and disabilities subclasses.

SECONDARY OUTCOMES:
the active ROM | baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The maximal active ROMs of the affected shoulder will be measured using a goniometer under the guidelines of the American Academy of Orthopedic Surgeons. These measurements included abduction in the frontal plane, forward flexion, internal rotation, and external rotation with the arm at 0 degrees of abduction.
Change of the Shoulder Disability Questionnaire (SDQ) | baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The SDQ is a symptoms-related questionnaire containing 16 items describing common situations that may induce symptoms in patients with shoulder disorders. By responding 'yes', 'no', or 'not applicable', the final score is obtained by dividing the number of positively scored items by the total number of applicable items and then multiplying this number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst situation).
Change of 36-item Short-Form Health Survey (SF-36) | baseline and at 4 weeks and 12 weeks after the beginning of the treatment.
  The SF-36 is a 36-item questionnaire that evaluates the quality of life. It is composed of 8 subscales: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale has a score range of 0 to 100, with a higher score indicating better health status.Patient's evaluation of the treatment effect. Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=1, effective=2, not effective=3, worse=4, much worse=5).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan